CLINICAL TRIAL: NCT01478867
Title: Phase 0 Monitoring of Gluten-free Diet Compliance in Celiac Patients by Assessment of Gliadin 33-mer Equivalent Epitopes in Feces
Brief Title: Detection of Immunotoxic Gluten Peptides in Feces
Acronym: CELIQK2
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Collaborators: Instituto Hispalense de Pediatría, Seville, Spain (Unknown)
Responsible Party: Principal Investigator, Carolina Sousa Martin, Principal Investigator, University of Seville
Other Study IDs: CELIQK2
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Celiac Disease
Keywords: celiac disease; gluten-free diet; gluten peptides; feces
MeSH Terms: conditions — Celiac Disease | interventions — Defecation; Diet, Gluten-Free

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Celiac patients
  Interventions: Other: Detection of gluten in feces

INTERVENTIONS:
Other: Detection of gluten in feces — Detection of Gluten in Feces
  Other Names: Gluten-free diet; Celiac patients

SUMMARY:
The purpose of this study is to monitor of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces.

DETAILED DESCRIPTION:
Certain immunotoxic peptides from gluten are resistant to gastrointestinal digestion and can interact with celiac patient factors to trigger immunological response. Gluten-free diet (GFD) is the only effective treatment for celiac disease (CD) and its compliance should be monitored to avoid accumulative damage. However, practical methods to monitor diet compliance and to detect the origin of an outbreak of celiac clinical symptoms are not available.

This study assesses the capacity to determine the gluten ingestion, and to monitor the GFD compliance in celiac patients by detection of gluten and gliadin 33-mer equivalent peptidic epitopes in human feces.

ELIGIBILITY:
Inclusion Criteria:

* Celiac patient
* 1-12 years old
* Written informed consent

Exclusion Criteria:

* Known inflammatory bowel diseases
* Participation in any other studies involving investigational concomitantly or within two weeks prior to entry into the study and during the course of the study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Celiac patients, 1-12 years old
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-04; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Monitoring of gluten-free diet compliance in celiac patients | April-July 2011 (3 months)
  Usual gluten diet for celiac (home diet not modified for this trial)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Sousa, Professor, Principal Investigator — University of Seville, Spain
Locations (1):
- Department of Microbiology and Parasitology, Faculty of Pharmacy, University of Seville, Seville, Seville, Spain

REFERENCES:
- [Background] Moron B, Cebolla A, Manyani H, Alvarez-Maqueda M, Megias M, Thomas Mdel C, Lopez MC, Sousa C. Sensitive detection of cereal fractions that are toxic to celiac disease patients by using monoclonal antibodies to a main immunogenic wheat peptide. Am J Clin Nutr. 2008 Feb;87(2):405-14. doi: 10.1093/ajcn/87.2.405. PMID 18258632
- [Background] Moron B, Bethune MT, Comino I, Manyani H, Ferragud M, Lopez MC, Cebolla A, Khosla C, Sousa C. Toward the assessment of food toxicity for celiac patients: characterization of monoclonal antibodies to a main immunogenic gluten peptide. PLoS One. 2008 May 28;3(5):e2294. doi: 10.1371/journal.pone.0002294. PMID 18509534
- [Background] Hausch F, Shan L, Santiago NA, Gray GM, Khosla C. Intestinal digestive resistance of immunodominant gliadin peptides. Am J Physiol Gastrointest Liver Physiol. 2002 Oct;283(4):G996-G1003. doi: 10.1152/ajpgi.00136.2002. PMID 12223360
- [Background] Shan L, Molberg O, Parrot I, Hausch F, Filiz F, Gray GM, Sollid LM, Khosla C. Structural basis for gluten intolerance in celiac sprue. Science. 2002 Sep 27;297(5590):2275-9. doi: 10.1126/science.1074129. PMID 12351792
- [Derived] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271